CLINICAL TRIAL: NCT04500561
Title: YY-20394 Combined With GEMOX in the Treatment of Patients With Relapsed and/or Refractory Diffuse Large B-cell Lymphoma With a Single Arm, Open, Multicentrized Phase 1b/2 Clinical Trial
Brief Title: YY-20394 、GEMOX Treatment Diffuse Large B-cell Lymphoma Single Arm, Open, Multicentrized Phase 1b/2 Clinical Trial
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YY-20394-008
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Gemcitabine; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: YY-20394 combined with GEMOX was used as a cycle for 21 days. The dose of YY-20394 was 80mg/ day as recommended in phase 2, and the dose of GEMOX was treated according to clinical standards
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YY-20394 (Experimental): YY-20394 tablets will be given daily for 21 days in 21-day cycles until there appears evidence of progressive disease, intolerable toxicity, or the subject discontinues from the study treatment for other reasons
  Interventions: Drug: YY-20394

INTERVENTIONS:
Drug: YY-20394 — Yy-20394 combined with Gemcitabine and Oxaliplatin was used as a cycle for 21 days. The dose of YY-20394 was 80mg/ day as recommended in phase 2, and the dose of Gemcitabine and Oxaliplatin was treated according to clinical standards.
  Other Names: Gemcitabine; Oxaliplatin

SUMMARY:
This study is a one-arm, open, multicenter phase 1b/2 clinical trial of YY-20394 combined with GEMOX second-line or above in patients with relapsed and/or refractory diffuse large B-cell lymphoma.

YY-20394 combined with GEMOX was used as a cycle for 21 days. The dose of YY-20394 was 80mg/ day as recommended in phase 2, and the dose of GEMOX was treated according to clinical standards.

DETAILED DESCRIPTION:
This study is a one-arm, open, multicenter phase 1b/2 clinical trial of YY-20394 combined with GEMOX second-line or above in patients with relapsed and/or refractory diffuse large B-cell lymphoma.

YY-20394 combined with GEMOX was used as a cycle for 21 days. The dose of YY-20394 was 80mg/ day as recommended in phase 2, and the dose of GEMOX was treated according to clinical standards.

The first six subjects of group to evaluate the safety of YY - 20394 joint GEMOX, if the joint treatment of 6 cases of subjects before, If YY-20394 and/or chemotherapy related 4 degrees of hematology toxicity or level 3 non hematologic toxicity were appearanced less than 2 cases, continued to dose of 80 mg/day, if more than 2 cases, YY-20394 doses dropped to 60 mg/day.

ELIGIBILITY:
Inclusion Criteria:

- Patients with recurrent and/or refractory diffuse large B-cell lymphoma confirmed histologically or cytologically; Progress after first-line or above systemic treatment (at least CD20 monoclonal antibody treatment); ECOG Performance Status (PS) grade 0 ~ 1; Expected survival ≥3 months; The patient has at least one measurable lesion conforming to the IWG2007 standard; Good organ function level:ANC≥1.0×109/L；PLT≥70×109/L；Hb≥80 g/L

;TBIL≤1.5×ULN； ALT和AST≤2.5×ULN；BUN/Urea和Cr≤1.5×ULN；LVEF≥50%； The Fridericia method corrected the QT interval (QTcF) for males < 450 ms and females < 470 ms.

From the end of any previous anti-tumor therapy (including radiotherapy, chemotherapy, hormone therapy, surgery or molecular targeted therapy) to the washout period of this study ≥4 weeks; Did not participate in the clinical trial as a subject within 1 month before the trial; According to the researcher's judgment, it can comply with the experimental protocol; Volunteer to participate in this clinical trial, understand the study procedures and be able to sign the informed consent in person.

Exclusion Criteria:

* Those who have used PI3K as the target of anti-tumor drug progression (except those who cannot tolerate out of the group); Any other anti-tumor therapy within 4 weeks; The presence of a third interstitial effusion that cannot be controlled by drainage or other methods (such as massive pleural and ascites); Use of steroid hormone dosage (equivalent amount of prednisone) greater than 20mg/ day within 4 weeks, and continuous use for more than 14 days; Unable to swallow, chronic diarrhea and intestinal obstruction, existing multiple factors affecting drug intake and absorption; Unable to suspend medications that may prolong QT interval during the study (e.g., antiarrhythmic agents); Having lympoma with central nervous system (CNS) invasion; Allergic constitution, or known anaphylaxis to any component of this product; Having active viral, bacterial or fungal infection requiring treatment (e.g., pneumonia); Uncontrolled diabetes, pulmonary fibrosis, acute pulmonary disease, interstitial lung disease, or liver failure; Patients with HBV, HCV infection (defined as HbsAg and/or HbcAb positive and HBV DNA copy number ≥1×104 copy number /ml or ≥2000 IU/ml) or acute or chronic active hepatitis C; Medical history of immunodeficiency, including HIV testing positive, or having other acquired or congenital immunodeficiency disease, or history of organ transplantation or allogeneic bone marrow transplantation; Having received autologous hematopoietic stem cell transplantation within 90 days prior to the first dose in this study; Any cardiac disease, including (1) angina pectoris; (2) arrhythmia requiring drug therapy or of clinical significance; (3) myocardial infarction; (4) heart failure; (5) any other cardiac disease that is judged by investigators as not suitable to participate in this trial; Pregnant or lactating women or baseline pregnancy testing positive for fertile women; Concomitant diseases (such as serious hypertension, diabetes mellitus, thyroid disease) seriously hazardous to patient's safety or completion of study as judged by the investigator; Having other primary malignancy in recent 5 years;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-08-20 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
objective remission rate | with in 42 days after the first dos
  Response will be determined by the revised International Working Group (IWG 2007) efficacy evaluation criteria

SECONDARY OUTCOMES:
disease control rate | with in 42 days after the first dos
  Response will be determined by the revised International Working Group (IWG 2007) efficacy evaluation criteria
Progression Free Survival | with in 42 days after the first dos
  Response will be determined by the revised International Working Group (IWG 2007) efficacy evaluation criteria
drug safety | one and half a year
  Adverse events evaluated by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Li, PHD, Principal Investigator — Cancer Prevention center affiliated to Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun P, Cen H, Yang H, Huang R, Cai Z, Gu X, Bao H, Xu Z, Xu Z, Li ZM. PI3Kdelta inhibitor linperlisib combined with gemcitabine and oxaliplatin for relapsed or refractory diffuse large B-cell lymphoma: a multicenter, single-arm phase Ib/II trial. Cancer Cell Int. 2025 Feb 8;25(1):39. doi: 10.1186/s12935-025-03669-2. PMID 39923042